CLINICAL TRIAL: NCT03200535
Title: Comparison of Outreach Methods to Encourage Enrollment in Diabetes Prevention and Weight Management Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Emily Schroeder, Investigator, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CO-17-2437
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: PreDiabetes; Obesity
MeSH Terms: conditions — Prediabetic State; Obesity

STUDY DESIGN:
Intervention Model Description: Individuals with a body mass index between 25 and 30 are randomized 1:1 to the Usual Care or EHR Gap arms. Individuals with a body mass index >=30 are randomized to all 4 arms, with n=1000 for the Personalized Outreach arm and 1:1:1 for the other three arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care (No Intervention): Usual care
- Electronic health record "gaps" (Active Comparator): Gaps will appear in the electronic health record and patient portal in order to prompt referral by provider or patient
  Interventions: Other: EHR gaps
- Bulk outreach (Active Comparator): Gaps will appear in the electronic health record and patient portal in order to prompt referral by provider or patient; in addition a bulk letter or email will be sent
  Interventions: Other: EHR gaps; Other: Bulk outreach
- Personalized outreach (Active Comparator): Gaps will appear in the electronic health record and patient portal in order to prompt referral by provider or patient; in addition a bulk letter or email will be sent and patients will receive a personalized call by a registered dietitian
  Interventions: Other: EHR gaps; Other: Bulk outreach; Other: Dietician call

INTERVENTIONS:
Other: EHR gaps — Gaps will appear in the electronic health record and patient portal in order to prompt referral by provider or patient
  Arms: Bulk outreach; Electronic health record "gaps"; Personalized outreach
Other: Bulk outreach — A bulk letter or email will be sent
  Arms: Bulk outreach; Personalized outreach
Other: Dietician call — Patients will receive a personalized call by a registered dietitian
  Arms: Personalized outreach

SUMMARY:
Individuals with prediabetes are at increased risk for developing diabetes. Higher hemoglobin A1c's (6.1-6.4%) are associated with a high risk of developing diabetes. It is known that programs such weight management classes and one-on-one counseling with registered dieticians can lead to weight loss and decrease the risk of diabetes. However, engagement of Kaiser Permanente Colorado members in these activities is low. The purpose of this study is to determine which of three outreach methods is most effective in increasing engagement in these activities.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Member
* Age 18-75
* Prediabetes
* BMI >= 25
* A1c 6.1-6.4%
* No dietitian visit within the past 3 years

Exclusion Criteria:

- Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6588 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Schroeder, MD, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Coloado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Electronic Health Record "Gaps" | Bulk Outreach | Personalized Outreach
Started | 1863 | 1863 | 1862 | 1000
Completed | 1863 | 1863 | 1862 | 1000
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Electronic Health Record "Gaps" | Bulk Outreach | Personalized Outreach | Total
Number analyzed (Participants) | 1863 | 1863 | 1862 | 1000 | 6588
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.9) | 58.2 (11.0) | 58.0 (11.1) | 58.3 (10.9) | 58.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 17 participants had missing data on gender
  Participants
    number analyzed (Participants) | 1857 | 1856 | 1861 | 997 | 6571
    Female | 999 | 1023 | 990 | 544 | 3556
    Male | 858 | 833 | 871 | 453 | 3015
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.3 (5.6) | 36.3 (6.1) | 36.6 (5.9) | 36.4 (5.5) | 36.4 (5.8)
A1c [Mean (Standard Deviation); unit: %] | 6.3 (0.18) | 6.3 (0.18) | 6.3 (0.18) | 6.3 (0.18) | 6.3 (0.17)

OUTCOME MEASURES:

1. Primary Outcome: Enrollment in Diabetes Prevention or Weight Management Class (Online)
Description: Percent of individuals who have enrolled in online diabetes prevention or weight management classes (online) over a 4.5 month period
Time Frame: 4.5 months (6/26/2017-11/10/2017)
Population: Entire population was analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic Health Record "Gaps" | Bulk Outreach | Personalized Outreach
Number analyzed (Participants) | 1863 | 1863 | 1862 | 1000
Participants | 7 | 12 | 39 | 59
Statistical Analysis 1: Comparison: Usual Care vs Electronic Health Record "Gaps" vs Bulk Outreach vs Personalized Outreach; Test type: Superiority — Superiority analysis; p < 0.001, Chi-squared

2. Secondary Outcome: Enrollment in Diabetes Prevention or Weight Management Class (in Person)
Description: Percent of individuals who have enrolled in diabetes prevention or weight management class (in person) over a 4.5 month follow-up period
Time Frame: 4.5 months (6/26/2017-11/10/2017)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic Health Record "Gaps" | Bulk Outreach | Personalized Outreach
Number analyzed (Participants) | 1863 | 1863 | 1862 | 1000
Participants | 15 | 14 | 24 | 25
Statistical Analysis 1: Comparison: Usual Care vs Electronic Health Record "Gaps" vs Bulk Outreach vs Personalized Outreach; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 4.5 months (6/26/2017-11/10/2017)
Arm/Group | Usual Care | Electronic Health Record "Gaps" | Bulk Outreach | Personalized Outreach
All-Cause Mortality (participants affected / at risk) | 2/1863 | 2/1863 | 3/1862 | 1/1000
Serious Adverse Events (participants affected / at risk) | 0/1863 | 0/1863 | 0/1862 | 0/1000
Other Adverse Events (participants affected / at risk) | 0/1863 | 0/1863 | 0/1862 | 0/1000

LIMITATIONS AND CAVEATS:
We were unable to analyze the change in BMI and change in A1c due to the low number of individuals who enrolled in diabetes prevention classes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT03200535/Prot_SAP_000.pdf